CLINICAL TRIAL: NCT06965543
Title: Randomized Controlled Clinical Trial Evaluating the Effect of Endoscopic Pyloromyotomy Via Gastric POEM on Glycemic Control in Patients With Diabetes and Gastroparesis
Brief Title: G-POEM for Glycemic Control in Diabetic Gastroparesis
Acronym: DIAPOEM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: French Society of Digestive Endoscopy (Other)
Responsible Party: Principal Investigator, Antoine DEBOURDEAU, Medical doctor, French Society of Digestive Endoscopy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SFED-166
Record Dates: First submitted 2025-04-16; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Gastroparesis
Keywords: G-POEM (Gastric Per Oral Endoscopic Myotomy); Gastroparesis; diabetic gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: Immediate G-POEM (Experimental)
  Interventions: Procedure: Immediate G-POEM
- Delayed G-POEM : Standard Treatment Followed by G-POEM at 3 Months (Active Comparator)
  Interventions: Procedure: Delayed G-POEM

INTERVENTIONS:
Procedure: Immediate G-POEM — Gastric POEM (G-POEM) performed under general anesthesia. A submucosal tunnel will be created along the greater curvature of the stomach to access the pyloric muscle under endoscopic vision. The pylorus will be incised at two locations with a dual myotomy between the 5 and 8 o'clock positions on the clock face
  Arms: Experimental Group: Immediate G-POEM
Procedure: Delayed G-POEM — Participants will receive standard medical treatment, including prokinetic agents, antiemetics (ondansetron 8 mg twice daily), nutritional support, and dietary counseling. Laxative treatments will be prescribed as needed. After three months, participants will undergo G-POEM as described above
  Arms: Delayed G-POEM : Standard Treatment Followed by G-POEM at 3 Months

SUMMARY:
Gastroparesis, commonly caused by diabetes, affects 30-50% of diabetic individuals and complicates glycemic control due to its bidirectional relationship with blood glucose levels. Current treatments are often ineffective. G-POEM, a minimally invasive endoscopic technique, has demonstrated promising results in improving digestive symptoms, particularly in diabetic patients, with over 80% success. However, its impact on glycemic control has not yet been investigated, highlighting the need for further research.

DETAILED DESCRIPTION:
Gastroparesis is a condition characterized by delayed gastric emptying, resulting in various digestive symptoms. Diabetes is the leading global cause of gastroparesis. This complication affects approximately 30-50% of individuals with diabetes, typically appearing after many years of disease progression and frequently in the presence of other vascular complications. It is associated with autonomic neuropathy and hyperglycemia.

The bidirectional relationship between gastric emptying and blood glucose levels contributes to the complexity of diabetes management, increasing the risk of both postprandial hypoglycemia and delayed hyperglycemia. Existing treatments, including prokinetic and antiemetic medications, are often poorly tolerated and of limited efficacy.

G-POEM (Gastric Per Oral Endoscopic Myotomy) is an endoscopic technique designed to treat refractory gastroparesis by targeting pyloric muscle hypertonicity. This procedure has demonstrated favorable outcomes in approximately two-thirds of cases and presents a favorable safety profile. The diabetic population appears to benefit most from this intervention, with over 80% reporting symptom improvement. To date, no study has evaluated the impact of G-POEM on glycemic parameters in patients with diabetic gastroparesis. This clinical trial aims to address this knowledge gap.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 90 years;
* Diagnosed with diabetes for at least 5 years and be treated with optimized insulin therapy;
* Severe gastroparesis with gastric retention >20% at 4h (confirmed by scintigraphy);
* Failure of conventional gastroparesis treatment;
* Continuous glucose monitoring (CGM) in use or willingness to use during study
* Time in range (70-180 mg/dL) <70%

Exclusion Criteria:

* Are treated with an automated insulin therapy system (closed-loop);
* Have previously undergone gastric neurostimulation therapy with Enterra (Medtronic ©);
* Have been treated with erythromycin in the past three months;
* Do not provide informed consent;
* Are pregnant or breastfeeding during the study period;
* Are under legal guardianship;
* Have contraindications to the POEM procedure, including contraindications to anesthesia and/or active anticoagulation that cannot be paused;
* Have severe chronic constipation, defined by a Cleveland score >15 (Agachan et al., Dis Colon Rectum, 1996);
* Have a history of esophagogastric surgery (excluding anti-reflux surgery), including esophagogastric resection or any type of bariatric surgery;
* Have chronic intestinal pseudo-obstruction;
* Have a clinical suspicion of chronic mesenteric ischemia, indicated by severe malnutrition, postprandial pain, and signs of digestive atherosclerosis;
* Refuse to share CGM data via the Libre Link platform;
* Plan or undergo changes in antidiabetic therapy or insulin delivery systems during the study period;
* Are being treated with any gastric-emptying delaying agents, including GLP-1 receptor agonists;
* Are undergoing treatment with ascorbic acid during the study;
* Have not previously attempted therapy with at least one prokinetic drug;
* Are actively treated with opioids;
* Have had prior pyloromyotomy or pyloroplasty;
* Have known eosinophilic gastroenteritis;
* Have an organic obstruction of the pylorus or intestinal tract (e.g., fibrotic stenosis);
* Have a severe coagulopathy;
* Have esophageal or gastric varices and/or portal hypertension gastropathy;
* Have decompensated liver cirrhosis (Child B or Child C);
* Have an active gastroduodenal ulcer;
* Have active cancer or precancerous conditions of the stomach or duodenum (dysplasia, gastric cancer, GIST).
* Have a known medical condition that, in the investigator's opinion, could interfere with the study protocol;
* Have experienced diabetic ketoacidosis requiring hospitalization within six months prior to enrollment;
* Have had a severe hypoglycemic episode requiring hospitalization within six months prior to enrollment.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of time spent in target glycemic range >10% | 3 months after randomization
  Proportion of time in the glycemic range 70-180 mg/dL calculated from CGM data over 14 days preceding the 3-month time point

SECONDARY OUTCOMES:
HbA1c Level | 15 days, 3 months, and 6 months after randomization
  Glycated hemoglobin (HbA1c) level measured in blood samples
Time in Hypoglycemia (<70 mg/dL) | 15 days, 3 months, and 6 months after randomization
  Percentage of time spent with glucose values below 70 mg/dL, based on continuous glucose monitoring (CGM) data.
Time in Hypoglycemia (<54 mg/dL) | 15 days, 3 months, and 6 months after randomization
  Percentage of time spent with glucose values below 54 mg/dL, based on continuous glucose monitoring (CGM) data.
Time in Hyperglycemia (>180 mg/dL) | 15 days, 3 months, and 6 months after randomization
  Percentage of time spent with glucose values above 180 mg/dL, based on continuous glucose monitoring (CGM) data.
Time in Hyperglycemia (>250 mg/dL) | 15 days, 3 months, and 6 months after randomization
  Percentage of time spent with glucose values above 250 mg/dL, based on continuous glucose monitoring (CGM) data.
Mean Glucose Level (mg/dL) | 15 days, 3 months, and 6 months after randomization
  Mean glucose level recorded by CGM over the specified time period.
Coefficient of Variation (CV) of Glucose (%) | 15 days, 3 months, and 6 months after randomization
  Coefficient of variation of glucose levels measured by CGM.
Gastric Emptying Assessment | 15 days, 3 months, and 6 months
  Evaluation of gastric motility via scintigraphy to measure gastric retention at 1h, 2h, and 4h post-standardized meal, performed at each follow-up time point (15 days, 3 months, and 6 months).
Fundic Accommodation Ratio | 15 days, 3 months, and 6 months
  Calculation of fundic accommodation using the ratio of T0 proximal activity to T0 total activity as per Orthey et al.
Gastroparesis Symptom Severity (GCSI Score) | 15 days, 3 months, and 6 months
  Gastroparesis symptoms assessed with the Gastroparesis Cardinal Symptom Index (GCSI), a validated questionnaire with a scale ranging from 0 to 5, where higher scores indicate more severe symptoms.
Severity of Upper GI Symptoms (PAGI-SYM Score) | 15 days, 3 months, and 6 months
  Patient-reported outcome measuring severity of upper GI symptoms using the PAGI-SYM questionnaire, a validated questionnaire with a scale from 0 to 5, where higher scores represent worse symptom severity.
Gastrointestinal Quality of Life (GIQLI Score) | 15 days, 3 months, and 6 months
  Quality of life related to gastrointestinal symptoms using the validated French version of the GIQLI scale.The total score ranges from 0 to 144, with higher scores indicating better quality of life.
Postprandial abdominal pain (VAS) | 15 days, 3 months, and 6 months
  Intensity of postprandial abdominal pain assessed using a visual analog scale (VAS) ranging from 0 (no pain) to 10 (worst imaginable pain).
Safety and Adverse Events | From inclusion to the end of the 6-month follow-up, over a total study duration of 36 months
  Number of participants experiencing serious or unexpected adverse events throughout the follow-up.